CLINICAL TRIAL: NCT04218188
Title: Evaluation of the Cell Detachment Ratio on pH-responsive Chitosan as a Prognostic Factor in Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201910061RINA
Record Dates: First submitted 2019-12-17; First posted 2020-01-06 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2019-12

CONDITIONS: Clinical Decision-Making; Early Detection of Cancer
Keywords: pH-responsive chitosan; Cancer stem-like cell; Cell detachment ratio; Prognostic factor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Biomaterial-based cell culture models have been gaining increasing attention as potential therapeutic strategies. The purpose of this project is to evaluate whether the cell detachment ratio on pH-responsive chitosan could be correlated with the overall survival in lung cancer patients. Through controllable cell-material interaction, this project has the intention to develop an alternative tool for both early diagnosis and accurate prognosis in cancer therapeutics.

ELIGIBILITY:
Inclusion Criteria:

* Lung cancer patient between 20-70 years old who need surgery for the resection of lung lesions.
* Willing to sign the consent form under the informed consent.

Exclusion Criteria:

* Vulnerable subjects included minors, prisoners, aborigines, pregnant women, people with mental disorders, students, and subordinates, etc.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At the discretion of the professional attending physician, the lung cancer patients who need to undergo resection of lung lesions.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-01-05 (Actual); Primary Completion 2020-11-17 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
The correlation between the cell detachment ratio and the overall survival | 5-year follow-up after tumor resection
  The purpose of this project is to evaluate whether the cell detachment ratio on pH-responsive chitosan could be correlated with the overall survival in lung cancer patients, hence serve as a prognostic factor for therapeutic strategies. The patient's information required for meta-analysis will be retrieved from medical records, and the log-term follow-up will be conducted.

SECONDARY OUTCOMES:
The analyses of the detached cells by specific markers | About one week
  The isolated and purified patient-derived tumor cells will be characterized by the expression of surface markers using flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Tai-Horng Young, Ph.D., Principal Investigator — Department of Biomedical Engineering, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan